CLINICAL TRIAL: NCT04175717
Title: Is a Physiotherapy-led Follow-up Programme Feasible in Adult Critical Illness Survivors After Discharge Home: A Single-center Trial
Brief Title: Feasibility of a Physiotherapy-led Follow-up Programme in Adult Critical Illness Survivors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID pandemic
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Principal Investigator, Natalie Ott, Clinical specialist in intensive care physiotherapy, Kantonsspital Winterthur KSW
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT-follow-up-post-ICU
Record Dates: First submitted 2019-11-07; First posted 2019-11-25 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Post Intensive Care Unit Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- physiotherapy-led follow-up programme (Experimental)
  Interventions: Other: physiotherapy-led follow-up programme

INTERVENTIONS:
Other: physiotherapy-led follow-up programme — In this study arm, the participants will receive a nine weeks exercise programme and four education sessions. During the exercise programme, the patients will exercise twice per week under supervision and once by themselves. The supervised exercise sessions will consisted out of a combination of a cardiopulmonary and strength training and the unsupervised session will be an activity, which the participants like doing. Additionally, when the patient shows a reduced maximal inspiratory pressure (indication for a reduced diaphragm strength), the patient will also be ask to do an inspiratory muscle training at home. Furthermore, they will participate in education sessions, where they learn things about the intensive care unit, the post-intensive care syndrome, relaxation techniques and how to carry on with exercising.

SUMMARY:
Survivors of critical illness might suffer from ongoing physical, cognitive and emotional impairments after being discharged home. Furthermore, several studies have shown that these patients might have a need for ongoing support. However, up until now, it is not known what the optimal follow-up programme for survivor of critical illness after discharge home should look like or which exact patient population would benefit the most. Due to these reasons, it is important to further investigate, how these patients can be optimally supported to recover from their critical illness.

The primary aim of this study is to assess, whether a physiotherapy-led follow-up programme is feasible in adult survivors of critical illness after discharge home in the county hospital of Winterthur.

Furthermore, the investigators evaluate the influence of this physiotherapy-led follow-up programme on health related quality of life, exercise capacity, general muscle strength, inspiratory muscle strength, anxiety and depression.

All of the anticipated 20 patients will partake in the follow-up programme, which will consist out of a nine weeks exercise programme and four education sessions. During the exercise programme, the patients will exercise twice per week under supervision and once by themselves. The supervised exercise sessions will consist out of a combination of a cardiopulmonary and strength training and the unsupervised session will be a physical activity, which the participants like doing. Furthermore, they will participate in education sessions, where they learn things about the intensive care unit, the post-intensive care syndrome, relaxation techniques and how to carry on with exercising.

The whole study will last about ten months and forms a part of a master thesis.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent after being informed
* Adult patient (>18 years), who was treated in the ICU of the county hospital of Winterthur and who was ventilated for longer than 48 hours
* Patient, who received inpatient rehabilitation and then was discharged home

Exclusion Criteria:

* Head or spinal cord injury, leading to neurological deficits
* Receiving palliative care
* Fractures diminishing mobility
* Principal diagnosis of chronic obstructive pulmonary disease (COPD)
* Principal diagnosis of myocardial infarction, heart failure or reanimation
* Principal diagnosis of stroke or cerebral bleeding
* Previous diagnosis of dementia or cognitive impairment
* Inability of the participant to follow the procedures of the study, e.g. due to language problems, psychological disorders, etc.;
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
The number of participants, who have completed the nine weeks physiotherapy-led follow-up programme | 10 weeks
  As part of the feasibility assessment of this physiotherapy-led follow-up programme in the county hospital of Winterthur, it will be assessed, how many participants are able to complete the whole programme.

SECONDARY OUTCOMES:
Health related quality of life | 10 weeks
  Health related quality of life will be measured by the EQ-5D L5 self-complete paper version, which is a self-report questionnaire. Th questionnaire contains five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), with each five levels (no problems, slight problems, moderate problems, severe problems, and extreme problems). The participants rate themselves in these levels. Additionally, they are also asked to rate their health on a visual analog scale from 0 (worst health you can imagine) to 100 (best health you could imagine).
Exercise capacity | 10 weeks
  Exercise capacity will be evaluated by the six minute walking test, which is a self-paced walking test to assess submaximal functional exercise capacity. The result will tell us, how many meters the participant could walk in six minutes.
General muscle strength | 10 weeks
  General muscle strength will be measured by the hand grip test with a Jamar dynamometer. The results will be reported in kilograms.
Inspiratory muscle strength | 10 weeks
  Inspiratory muscle strength will be evaluated by the CareFusion micro RPM, which measures the maximal inspiratory pressure at the level of the mouth. The results will be reported in centimeter of water.
Anxiety and Depression | 10 weeks
  Levels of anxiety and depression will be assessed by the hospital anxiety and depression scale (HADS), which is a self-administered questionnaire. It contains 14 items (seven to assess anxiety levels und seven to assess depression levels). Each item can be scored from zero to three, leading to a maximal score of 21. The higher a participants scores, the more likely he is to suffer from anxiety or depression (or both).

CONTACTS AND LOCATIONS:
Overall Officials: Ott Natalie, Principal Investigator — Institut für Therapien und Rehabilitation, Kantonsspital Winterthur
Locations (1):
- Kantonsspital Winterthur, Winterthur, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Cuthbertson BH, Roughton S, Jenkinson D, Maclennan G, Vale L. Quality of life in the five years after intensive care: a cohort study. Crit Care. 2010;14(1):R6. doi: 10.1186/cc8848. Epub 2010 Jan 20. PMID 20089197
- [Background] Davydow DS, Gifford JM, Desai SV, Bienvenu OJ, Needham DM. Depression in general intensive care unit survivors: a systematic review. Intensive Care Med. 2009 May;35(5):796-809. doi: 10.1007/s00134-009-1396-5. Epub 2009 Jan 23. PMID 19165464
- [Background] Desai SV, Law TJ, Needham DM. Long-term complications of critical care. Crit Care Med. 2011 Feb;39(2):371-9. doi: 10.1097/CCM.0b013e3181fd66e5. PMID 20959786
- [Background] King J, O'Neill B, Ramsay P, Linden MA, Darweish Medniuk A, Outtrim J, Blackwood B. Identifying patients' support needs following critical illness: a scoping review of the qualitative literature. Crit Care. 2019 May 24;23(1):187. doi: 10.1186/s13054-019-2441-6. PMID 31126335
- [Background] Prinjha S, Field K, Rowan K. What patients think about ICU follow-up services: a qualitative study. Crit Care. 2009;13(2):R46. doi: 10.1186/cc7769. Epub 2009 Apr 1. PMID 19338653
- [Background] Taito S, Yamauchi K, Tsujimoto Y, Banno M, Tsujimoto H, Kataoka Y. Does enhanced physical rehabilitation following intensive care unit discharge improve outcomes in patients who received mechanical ventilation? A systematic review and meta-analysis. BMJ Open. 2019 Jun 9;9(6):e026075. doi: 10.1136/bmjopen-2018-026075. PMID 31182443